CLINICAL TRIAL: NCT06225193
Title: Exploratory Analysis of Enhanced Liver Function (ELF) Test to Detect Early Fatty Liver in High Risk Population
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 022.HEP.2023.D
Record Dates: First submitted 2023-11-13; First posted 2024-01-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this initial investigator-initiated retrospective study, aim to analyze the enhanced liver fibrosis (ELF) scores in this high-risk population for NAFLD/nonalcoholic steatohepatitis(NASH)-related fibrosis. Study define 'high-risk' to include metabolic syndrome, which can be further defined by an atherosclerotic cardiovascular disease (ASCVD) score >7.5, any diagnosis of hyperlipidemia, history of coronary artery disease, history of heart failure, hypertension and/or type 2 diabetes. Study would also like to compare the performance of this score with historical methods of fibrosis assessment, where applicable, including vibration-controlled transient elastography, magnetic resonance elastography, blood markers and liver biopsy. Study will assess the impact of ELF scores on predicting liver events in the time, have used it and determine if diet, lifestyle changes and/or pharmacotherapy will improve serial ELF scores. Will also seek to understand how ELF scores are distributed in our community.

DETAILED DESCRIPTION:
Methodist Health System consists of nine hospitals and over one hundred clinics that serve 7% to 10% of patients in the Dallas metropolitan. In November 2021, adopted the use of ELF tests in patients who had risk factors for NAFLD/NASH based on abnormal liver enzymes, metabolic risk factors, and evidence of hepatosteatosis on imaging. There is a knowledge gap in the literature when it comes to ELF scores in our population and the data we collect in this study will contribute to filling that knowledge gap.

Historically, assessment of fibrosis has been accomplished with FibroScan,elastography or liver biopsy. However, these tests are not widely available in most clinics, and can be invasive and costly. At present, the two primary inexpensive and non-invasive alternatives are the fibrosis-4 (FIB-4) and ELF scores, which employ algorithms that utilize routine lab draws. While a low FIB-4 score has a negative predictive value of 90% for advanced fibrosis, it does not provide a risk assessment of liver-related events. For this reason, the study explore the newer ELF serum test as a non-invasive, more affordable and available means to detect patients with developing fibrosis and as a predictor of liver-related outcomes that could be easily used in a primary care setting. This will better risk-stratify this patient population at the primary care level, without need for invasive and expensive testing, and will guide appropriate referrals to Hepatology.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* NAFLD/NASH and non-NAFLD/NASH patients who have had an assessment with ELF score at Methodist Dallas Medical Center from November 2021 to December 2023.

Exclusion Criteria:

* Patients with incomplete data and those lost to follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 18 years of age, NAFLD/NASH and non-NAFLD/NASH who have assessed with ELF score at Methodist Dallas Medical Center from November 2021 to December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Enhanced Liver Fibrosis (ELF )scores | 6 months
  Will measure the ELF scores-Reference range 7.14-9.55, the lowest value means better and highest value would mean worst
Instances of hospital admission for ascites, edema/anasarca, portal hypertensive-related bleeding or encephalopathy | 6 months
  Number of hospital admissions for ascites, edema/anasarca, portal hypertensive-related bleeding or encephalopathy
Demographics | 6 months
  age (years), gender (male/female), race (Caucasian, Black, Hispanic, Asian, Other)
Instances of comorbidities | 6 months
  Patients with hypertension(HTN), Hypersensitivity Lung Disease(HLD), Coronary Artery Disease(CAD),Heart Failure( HF), Atherosclerotic cardiovascular disease (ASCVD), Type 2 Diabetes Mellitus(T2DM) as comorbidities

SECONDARY OUTCOMES:
Abnormalities in Liver ultrasound (U/S) findings | 6 months
  rate of liver damage
Abnormalities in Liver biopsy results | 6 months
  Rate of cancerous cells in liver

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, MD, Principal Investigator — Methodist Midlothian Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No